CLINICAL TRIAL: NCT03716518
Title: Effect of TCM-TSKSR on Completion Rates of Chemotherapy in Patients With Stage II & III Colon Cancer: A Randomized Placebo-Controlled Clinical Trial
Brief Title: Herbal Treatment to Improve Chemotherapy Delivery
Acronym: HATCHED
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing University of Chinese Medicine (Other); Peking University Third Hospital (Other); Beijing Chao Yang Hospital (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Shanghai Zhongshan Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Tianjin Union Medical Center (Other); Henan Provincial People's Hospital (Other); Zhengzhou Hospital of Traditional Chinese Medicine (Other); Peking University Cancer Hospital & Institute (Other); Chongqing University Cancer Hospital (Other); Civil Aviation General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017YFC1700604
Record Dates: First submitted 2018-10-14; First posted 2018-10-23 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-11

CONDITIONS: Colon Cancer
Keywords: Colon Cancer; Traditional Chinese Medicine; Adverse Effect of Chemotherapy; Chemotherapy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM group (Experimental): Tonifying Spleen and Kidney Sequential Regimen(TSKSR) will be prescribed to the participants in each course of chemotherapy.
  Interventions: Drug: Tonifying Spleen and Kidney Sequential Regimen
- Placebo group (Placebo Comparator): Placebo of Tonifying Spleen and Kidney Sequential Regimen(TSKSR)similar in color,smell and texture with TSKSR will be prescribed to participants in each course of chemotherapy.
  Interventions: Drug: Placebo of 'Tonifying Spleen and Kidney Sequential Regimen

INTERVENTIONS:
Drug: Tonifying Spleen and Kidney Sequential Regimen — TSKSR will be given to the participants as follows:Liu-jun-an-wei Granule,1 pack each time,twice a day,PO,from 0 to 6th day of chemotherapy and Qi-tu-er-zhi Granule,1 pack each time,twice a day,PO,from 7th to 20th day of chemotherapy.
  Other Names: TSKSR
  Arms: TCM group
Drug: Placebo of 'Tonifying Spleen and Kidney Sequential Regimen — Placebo of TCM-TSKSR will be given to the participants as follows:placebo of Liu-jun-an-wei Granule,1 pack each time,twice a day,PO,from 0 to 6th day of chemotherapy and placebo of Qi-tu-er-zhi Granule,1 pack each time,twice a day,from 7th to 20th day of chemotherapy.
  Other Names: Placebo of TSKSR
  Arms: Placebo group

SUMMARY:
This study is designed to:(1) determine the efficacy of Traditional Chinese Medicine (TCM) 'Tonifying Spleen and Kidney Sequential Regimen' (TSKSR) in improving the completion rate of 8-cycle CapeOX chemotherapy in patients with stage II (high-risk)& III colon cancer;(2) evaluate the efficacy of the TCM-TSKSR on adverse events of CapeOX chemotherapy and it's impact on patients' quality of life (QoL).A randomized,double-blinded,placebo-controlled clinical trial including seven centers will be conducted in Mainland China.The study will enroll patients with stage II (high-risk)& III colon cancer who have completed radical surgery and are going to receive CapeOX chemotherapy.All participants will receive chemotherapy as prescribed by their treating physicians and be randomly assigned to either concurrent use of TCM-TSKSR or placebo.

DETAILED DESCRIPTION:
CapeOX chemotherapy is a combination therapy of Oxaliplatin 130mg/m^2 IV on 1st day and Capecitabine 1000mg/m^2 PO twice daily from 1th day to 14th day,21 days for each course of treatment.Adverse effects of chemotherapy,such as myelosuppression and gastrointestinal reactions,may lead to dose reductions,treatment delays or even discontinuation among cancer patients. According to IDEA study,the completion rate of 8-cycle CapeOX chemotherapy in colorectal cancer patients is 64%,which means that nearly 4 in 10 patients could not complete adjuvant chemotherapy as planned,which may negatively impact patients' survival outcomes.Some prior studies have shown that TCM can improve patients' symptom control and QoL during adjuvant chemotherapy,which may further improve the completion of adjuvant chemotherapy. However,there is a lack of definitive evidence to evaluate the effects of TCM in stage II(high-risk)& III colon cancer patients who receive adjuvant chemotherapy after radical surgery.The study will be conducted between 2018 and 2021.Four hundred participants will be enrolled and randomly assigned to either the experimental group or the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pathological diagnosis of colon cancer; no residual tumor at the resection margin.
* tumor-node-metastasis(TNM)Stage II (high-risk)or III colon cancer according to 8th edition of American Joint Committee on Cancer(AJCC)Staging Manual. High-risk stage II disease is characterized by at least one of the following:

  1. T4 tumor,
  2. inadequately sampled nodes (<12 lymph nodes),
  3. clinical presentation with bowel obstruction or perforation,
  4. poorly differentiated histology ,exclusive of those cancers that are High degree of microsatellite instability(MSI-H),
  5. lymphovascular invasion,perineural invasion(PNI).
* Underwent radical surgery no more than six weeks ago and plan to start chemotherapy.
* Have not been enrolled in other therapeutic clinical trials within the near 30 days.
* Age between 18 to 75 years; All genders; Eastern Cooperative Oncology Group - performance status(ECOG-PS)from 0 to 2; Women who are pregnant, lactating or of reproductive age are not eligible, while those of reproductive age using secure contraceptives are eligible.
* No history of previous malignancy other than adequately treated in situ carcinoma of the uterine cervix or basal or squamous cell carcinoma of the skin, unless there has been a disease-free interval of at least 5 years.
* Laboratory testing: blood routine examination: WBC≥3.5×109/L，NEUT≥1.5×109/L,PLT≥100×109/L,HGB≥90g/L;biochemical tests:TBIL≤1.5×ULN,AST(SGOT),ALT(SGPT)≤2.5×ULN,Scr≤1.5×ULN;CEA after surgery was normal.
* Consented.
* Agree not to be enrolled in other interventional studies during the research.

Exclusion Criteria:

* Patients not suitable for chemotherapy of CapeOX ,which will be determined by the investigator or the attending physician.
* Clinically relevant cardiovascular and/or cerebrovascular disease,active hepatitis,severe abnormalities in liver/ renal function tests.
* Known allergy to any of the components of study drug.
* Those who cannot take the study drug orally because of bowel obstruction and/or require for peripheral vein nutrition.
* Malabsorption or diseases that affect the absorption.
* Unstable situations or situations that may endanger the safety of patients and their compliance, such as severe mental illness,schizophrenia.
* Colostomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Completion Rate of 8-cycle Adjuvant Chemotherapy | 6months
  Completion Rate of 8-cycle Adjuvant Chemotherapy=number of participants completing 8-cycle adjuvant chemotherapy/number of participants randomized to each group*100%

SECONDARY OUTCOMES:
Completion Rate of Adjuvant Chemotherapy of Each Participant | 6months
  Completion Rate of Adjuvant Chemotherapy of Each Participant=number of the last courses of chemotherapy/8*100%
Completion Rate of 4-cycle Adjuvant Chemotherapy | 3months
  Completion Rate of 4-cycle Adjuvant Chemotherapy=number of participants completing 4-cycle adjuvant chemotherapy/number of participants randomized to each group*100%
Time to Treatment Failure,TTF | 6months
  TTF is the period from randomization to the earliest day of an event such as withdrawal from protocol treatment for any reasons, patients refusal and loss to follow-up.
Relative Dose Intensity (RDI) of Adjuvant Chemotherapy | 6months
  Relative dose intensity (RDI) (%) = (actual dose/ initial dose of adjuvant chemotherapy) × 100%
Proportion of Modifications of Time | 6months
  Proportion of Modifications of Time=number of participants delaying chemotherapy /number of participants randomized to each group*100%.Delay is defined as ≥7days because of adverse event,such as weakness, myelosuppression, gastrointestinal reactions and other toxicity,except for administrative issues related to hospitalization.
Time of Dose Reductions of Adjuvant Chemotherapy for the First Time | 6months
  It is the period from randomization to when a chemo-induced grade 3-4 granulocytopenia and/or a chemo-induced grade 2 thrombocytopenia is observed in participants for the first time,in which case,the dose of both Oxaliplatin and Capecitabine will be reduced by 25% of planned dosage.
Time of Dose Reductions of Adjuvant Chemotherapy for the Second Time | 6months
  It is the period from randomization to when a chemo-induced grade 3-4 granulocytopenia and/or a chemo-induced grade 2 thrombocytopenia is observed in participants for the second time,in which case,the dose of both Oxaliplatin and Capecitabine will be reduced by 50% of planned dosage.
Proportion of Salvage Treatment | 6months
  Proportion of Salvage Treatment=Number of participants receiving salvage treatment/Number of participants randomized to each group*100%.
Incidence of a Chemo-induced Grade 3-4 Nausea/Vomiting | 6 months
Incidence of a Chemo-induced Grade 2 Diarrhea | 6 months
Changes of Participants' ESAS Score | 6 months
  Edmonton Symptom Assessment Scale(ESAS) score will be used to evaluate the change of participants' QoL during adjuvant chemotherapy.ESAS has 9 items designed to assess the severity of commonly reported symptoms experienced by cancer patients,including pain, fatigue, drowsiness, nausea, dyspnea, depression, anxiety, well-being, and loss of appetite.Each items ranges from 0 to 10.
Changes of Participants' FACT-C Score | 6months
  Functional Assessment of Cancer Therapy-Colorectal (FACT-C) score will be used to evaluate the change of participants' QoL during adjuvant chemotherapy.The FACT-C consists of 36 items,in four domains of well-being (physical,emotional,social,and functional),on a scale of 0 to 4.
Changes of TCM Symptoms Score | 6months
  Based on a prior expert consensus,11 TCM symptoms were considered to be the most common symptoms during CapeOX chemotherapy,including vomiting, numbness, diarrhea, constipation, sensation of chill, nocturia, forgetfulness, spontaneous sweating, night sweats, dry mouth and canker sores, each of which ranges from 0 to 10.
Changes of Spleen Deficiency Scale Score | 6months
  Based on prior researches,the investigator designed Spleen Deficiency Scale,which includes 8 items involving appetite,abdominal distension and so on.Each question ranges from 1 to 5.
Changes of Kidney Deficiency Scale Score | 6months
  Based on prior researches,the investigator designed Kidney Deficiency Scale, which includes 8 items involving soreness of waist, tinnitus, and so on. Each question ranged from 1 to 5.
Incidence of AEs | 6months
  Adverse effects(AEs) includes abnormal results of blood/urine/stool routine examination, liver/renal function test and electrocardiograms.
Incidence of SAEs | 6months
  Serious Adverse effects(SAEs) includes abnormal results of blood/urine/stool routine examination, liver/renal function test and electrocardiograms.

CONTACTS AND LOCATIONS:
Overall Officials: Yufei Yang, M.D., Principal Investigator — Xi-Yuan Hospital, China Academy of Chinese Medical Sciences
Locations (12):
- China (12):
  - Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - Civil Aviation General Hospital, Beijing, Beijing Municipality
  - Oncology Department of Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangdong, Guangzhou
  - The Third People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhengzhou Hospital of Traditional Chinese Medicine, Zhengzhou, Henan
  - Jiangsu Province Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Tianjin Union Medical Center, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang T, Fei YT, Xu Y, Sun LY, He B, Yan SH, Tang M, Yan YZ, Mao J, Yang YF. Effect of Jianpi Bushen Sequential Formula on Adjuvant Chemotherapy of Colon Cancer: Study Protocol for a Randomized Controlled Trial. Chin J Integr Med. 2021 Dec;27(12):891-895. doi: 10.1007/s11655-021-3448-9. Epub 2021 Aug 25. PMID 34432206